CLINICAL TRIAL: NCT05104489
Title: A Phase I/II, Placebo-Controlled, Randomized, Double-Blind, Dose-Finding Study to Evaluate the Safety, Tolerability, and Immunogenicity of AdimrSC-2f Vaccine in Healthy Adults
Brief Title: Dose-finding Study for AdimrSC-2f Vaccine
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Adimmune Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ADPCT21013I
Record Dates: First submitted 2021-10-04; First posted 2021-11-03 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Low Dose (Experimental): 50 mcg of antigen with 250 mcg of Al(OH)3
  Interventions: Biological: AdimrSC-2f
- Median Dose (Experimental): 100 mcg of antigen with 250 mcg of Al(OH)3
  Interventions: Biological: AdimrSC-2f
- High Dose (Experimental): 100 mcg of antigen with 500 mcg of Al(OH)3
  Interventions: Biological: AdimrSC-2f
- Placebo (Placebo Comparator): 250 mcg of Al(OH)3
  Interventions: Biological: AdimrSC-2f

INTERVENTIONS:
Biological: AdimrSC-2f — IM injection

SUMMARY:
AdimrSC-2f is a subunit protein-based vaccine produced using the baculovirus insect cells manufacturing process to prevent Coronavirus disease 2019 (COVID-19). The primary goal of this Phase I/II study is to evaluate the vaccine safety and immunogenicity of AdimrSC-2f in healthy adult individuals, as compared to placebo.

DETAILED DESCRIPTION:
This will be a Phase I/II, placebo-controlled, randomized, double-blind within dose cohort, dose-finding study to evaluate the safety, tolerability, and immune response of AdimrSC-2f vaccine against severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) in healthy adults aged from 18 to 60. Two hundred forty (240) subjects will be sequentially enrolled from low dose to high dose cohort and then randomized into AdimrSC-2f vaccine group or matched placebo in a 3:1 ratio. Each enrolled subject will receive a total of 3 doses with 3-week apart by 0.5 mL intramuscular (IM) injection to the deltoid region of non-dominant arm preferably. All enrolled subjects will be follow their safety and immune response for six months.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged 18 to 60 years old (inclusive) at the time of informed consent who are in good general health in the opinion of the investigator.
2. At Screening Visit, subjects with a body mass index (BMI) > 18.5 kg/m2 or ≤ 30.0 kg/m2.
3. Subjects without known history of SARS-CoV-2 infection or known close contact with anyone with laboratory-confirmed SARS-CoV-2 infection or COVID-19 within 2 weeks prior to the first dosing.
4. Subjects are willing and able to give informed consent prior to any screening procedure conducting and to comply with study procedures.
5. Female subjects of childbearing potential (defined as any female who has experienced menarche and who is NOT surgically sterile [ie, hysterectomy, bilateral tubal ligation, or bilateral oophorectomy] or postmenopausal [defined as amenorrhea at least 12 consecutive months or documented plasma follicle-stimulating hormone level ≥40 milli-International unit (mIU)/mL]) must agree to be heterosexually inactive from at least 21 days prior to the Screening Visit and through 6 months (defined as 24 weeks) after the last dosing OR agree to consistently use any of the following methods of contraception from at least 21 days prior to the Screening Visit and through 6 months (defined as 24 weeks) after the last dosing:

   * Condoms (male or female) with spermicide (if acceptable in country)
   * Diaphragm with spermicide
   * Cervical cap with spermicide
   * Intrauterine device
   * Oral or patch contraceptives
   * Norplant®, Depo-Provera®, or other in country regulatory-approved contraceptive method that is designed to protect against pregnancy
   * Abstinence, as a form of contraception, is acceptable

Exclusion Criteria:

1. Subjects who are investigational site staff member directly involved in the conduct of the trial and their family members, site staff members otherwise supervised by the Investigator, or subjects who are Sponsor employees directly involved in the conduct of the trial.
2. Any ongoing severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.
3. Subject with positive serology test results for human immunodeficiency virus (HIV), hepatitis C virus (HCV) or hepatitis B virus (HBV) at the Screening Visit (V0).
4. Subject with positive test result for COVID-19 antigen rapid test at the Screen Visit or V1 prior to the 1st dosing.
5. Subject with influenza-like illness as defined by any of the following symptoms at the Screening Visit or before randomization: fever (tympanic temperature ≥ 38°C), dry cough, headache, fatigue, respiratory sputum production (phlegm), dysgeusia, anosmia, shortness of breath, muscle and joint pain, or sore throat.
6. Participation in other studies involving investigational drug(s) and/or device(s) within 90 days prior to the Screening Visit and/or during study participation.
7. Subject who has received any investigational coronavirus vaccine or has received any medications intended to prevent COVID-19 or plan simultaneous participation in another interventional study to prevent or treat COVID-19.
8. Subject with any following ongoing disease or medical history in medical chart or by verbal confirmation:

   * Diagnosis of malignancy not in remission for the past 3 years except non-melanoma skin cancer prior to the Screening Visit.
   * Chronic pulmonary disease, asthma or wheezing.
   * Chronic liver disease or suspected active hepatitis.
   * Clinically significant cardiovascular disease such as arrhythmia, coronary artery disease or heart failure.
   * Personal or family history of immune disorders, including systemic lupus erythematosus (SLE), rheumatoid arthritis, multiple sclerosis, inflammatory bowel disease, and Type 1 diabetes.
   * Any confirmed or suspected abnormal immune function, immunosuppressive, or immunodeficiency.
   * Personal or family history of Guillain-Barré Syndrome.
   * Bleeding diathesis or condition associated with prolonged bleeding.
   * History of anaphylaxis, urticarial or severe adverse reaction associated with a vaccine or AdimrSC-2f or aluminum.
   * Dermatologic conditions that could affect local solicited adverse event assessment per the investigator's opinion.
9. Subject who has any of the following prior medication histories:

   * Received any vaccine (live, inactivated, or bacterial) within 30 days prior to the Screening Visit.
   * Received any blood/plasma products or immunoglobulin within 90 days prior to the Screening Visit.
   * Received any systemic corticosteroids or steroids within 30 days prior to the first dosing. Topical, inhaled/nebulized, intra-articular, or nasal corticosteroid/ steroids are permitted.
   * Received treatment with immunosuppressive therapy, including cytotoxic agents, immunosupressants or system corticosteroids for organ transplant, cancer, or an autoimmune disease, or planned receipt for disease treatment during study period.
   * Used bronchodilator within 90 days prior to the Screening visit.
10. Subject with current use or history of chronic smoking (defined as ≥ 1 cigarette per day) in the medical chart or by verbal confirmation within 1 year prior to the Screening Visit.
11. Subject with the history of illegal substance use or alcohol abuse in the medical chart or by verbal confirmation within 2 years prior to the Screening Visit.
12. Female subject who is pregnant or lactating at the Screening Visit or Visit 1 or plan to be pregnant during the study period.
13. Subject who has donated ≥ 250 mL of blood product within 28 days prior to the Screening Visit or who plans to donate blood products during the study period.
14. Subject with levels of creatine phosphokinase outside of the reference range at the Screening Visit.
15. Subject who is not suitable to participate in this study as judged by the investigator.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 241 (Actual)
Dates: Start 2022-01-03 (Actual); Primary Completion 2022-12-29 (Actual); Study Completion 2023-07-26 (Actual)

PRIMARY OUTCOMES:
SARS-CoV-2 neutralizing antibody tiers | 21 days after the 3rd dosing
Incidence of adverse events and clinically significant changes in clinical and laboratory evaluations. | Day 1 to 24 weeks after the last dosing

SECONDARY OUTCOMES:
SARS-CoV-2 neutralizing antibody tiers | Day 1, Day 22, Day 43, 21 days after the last dosing, and 24 weeks after the last dosing
Number of subjects with SARS-CoV-2 infection | 21 days after the 3rd dosing to 24 weeks after the last dosing

CONTACTS AND LOCATIONS:
Locations (1):
- University Gadjah Mada Academic Hospital, Yogyakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No